CLINICAL TRIAL: NCT04528485
Title: The Effect of a Sea-safety Course on Mood, Mental Wellbeing and Inflammation
Brief Title: Sea Swimming for Treatment of Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Devon Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DPT0468 Sea Swimming
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sea swimming (Experimental): 8 sessions over 4 weeks of swimming-based activities in the sea
  Interventions: Other: Sea swimming

INTERVENTIONS:
Other: Sea swimming — 8 sessions of swimming activities in the sea

SUMMARY:
There is a developing evidence to suggest that open cold water swimming could have an impact on depression and anxiety:

* anecdotal reports of benefits to mental wellbeing as a result of regular open water bathing
* research suggesting exercise is as effective as medication and talking therapies in the treatment of depression
* ecotherapy (offering therapeutic intervention in nature) has a developing evidence base
* cold water may have an impact on the inflammatory system which has been linked to depression

The aim of this study is to recruit 10 people with mild to moderately severe depression to a sea swimming course, alongside their standard care. The course would involve two groups of 5, participating in eight sea sessions under the guidance and supervision of swim instructors and lifeguards.

The primary aim of the course is to determine the recruitment rate and compliance with the course.

The secondary aims of the course are to determine the impact on mental health through questionnaires for depression (PHQ9), anxiety (GAD7), functioning in daily life (WSAS). The inflammatory marker - C- reactive protein (CRP), will also be measured to monitor the inflammatory process in relation to psychological outcomes and the timeline of the course.

Participants will need to commit to two sessions a week. It is anticipated that participants will need to commit around 2 hours of their time to the study each week.

It would take around ten months from recruitment to follow-up. Participants would be able to leave the study at any time. Participants would engage in routine care alongside the course.

Sea swimming can be a dangerous activity but participants would be well supported, in small groups and would only sea swim in safe conditions. Participants will be asked to report any medical conditions to ensure they could not be adversely effected.

ELIGIBILITY:
Inclusion Criteria:

* Adults living in North Devon and able to attend the course.
* PHQ-9 score 5-19
* Able to swim two lengths of a 25m pool

Exclusion Criteria:

* Physical health problems that would make cold water immersion a risk including significant heart problems, inadequately treated high blood pressure e.g. new diagnosis not on stable medication, significantly reduced mobility.
* Experience of other mental health problems at a significant level
* Not able to swim or very anxious about getting into water
* Suicide risk
* Unable to speak English (as the sea swimming course will be conducted in English)
* Unable to consent due to lack of capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention of participants | 5 weeks
  The number of participants recruited and how many of them complete the course

SECONDARY OUTCOMES:
Effect of course on measures of anxiety | 5 weeks
  Comparison of GAD7 scores before the start and after completion of the intervention
Effect of course on measures of depression | 5 weeks
  Comparison of PHQ9 scores before the start and after completion of the intervention
Effect of course on measures of functioning | 5 weeks
  Comparison of WSAS scores before the start and after the completion of the intervention
Effect of course on inflammation | 5 weeks
  Comparison of CRP pre- and post-course

CONTACTS AND LOCATIONS:
Overall Officials: C Mark Harper, MBBS, Study Chair — Brighton and Sussex University Hospitals
Locations (1):
- Croyde Beach, Croyde, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beilin B, Shavit Y, Razumovsky J, Wolloch Y, Zeidel A, Bessler H. Effects of mild perioperative hypothermia on cellular immune responses. Anesthesiology. 1998 Nov;89(5):1133-40. doi: 10.1097/00000542-199811000-00013. PMID 9822001
- [Background] Bryleva EY, Keaton SA, Grit J, Madaj Z, Sauro-Nagendra A, Smart L, Halstead S, Achtyes E, Brundin L. The acute-phase mediator serum amyloid A is associated with symptoms of depression and fatigue. Acta Psychiatr Scand. 2017 May;135(5):409-418. doi: 10.1111/acps.12730. Epub 2017 Apr 4. PMID 28374419
- [Background] Canli T. Reconceptualizing major depressive disorder as an infectious disease. Biol Mood Anxiety Disord. 2014 Oct 21;4:10. doi: 10.1186/2045-5380-4-10. eCollection 2014. PMID 25364500
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] Denton, H. and Aranda K. The wellbeing benefits of sea swimming. Is it time to revisit the sea cure? Qualitative Research in Sport, Exercise and Health. 2019. pp. 1-17.
- [Background] Dugdill L, Graham RC, McNair F. Exercise referral: the public health panacea for physical activity promotion? A critical perspective of exercise referral schemes; their development and evaluation. Ergonomics. 2005 Sep 15-Nov 15;48(11-14):1390-410. doi: 10.1080/00140130500101544. PMID 16338708
- [Background] Foley R. Swimming in Ireland: Immersions in therapeutic blue space. Health Place. 2015 Sep;35:218-25. doi: 10.1016/j.healthplace.2014.09.015. PMID 25456012
- [Background] Gabay C, Kushner I. Acute-phase proteins and other systemic responses to inflammation. N Engl J Med. 1999 Feb 11;340(6):448-54. doi: 10.1056/NEJM199902113400607. No abstract available. PMID 9971870
- [Background] Hage FG, Szalai AJ. C-reactive protein gene polymorphisms, C-reactive protein blood levels, and cardiovascular disease risk. J Am Coll Cardiol. 2007 Sep 18;50(12):1115-22. doi: 10.1016/j.jacc.2007.06.012. Epub 2007 Sep 4. PMID 17868801
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Iacobucci G. NHS prescribed record number of antidepressants last year. BMJ. 2019 Mar 29;364:l1508. doi: 10.1136/bmj.l1508. No abstract available. PMID 30926584
- [Background] Jones A, Hillsdon M, Coombes E. Greenspace access, use, and physical activity: understanding the effects of area deprivation. Prev Med. 2009 Dec;49(6):500-5. doi: 10.1016/j.ypmed.2009.10.012. Epub 2009 Oct 24. PMID 19857513
- [Background] Maes M, Delange J, Ranjan R, Meltzer HY, Desnyder R, Cooremans W, Scharpe S. Acute phase proteins in schizophrenia, mania and major depression: modulation by psychotropic drugs. Psychiatry Res. 1997 Jan 15;66(1):1-11. doi: 10.1016/s0165-1781(96)02915-0. PMID 9061799
- [Background] Markanday A. Acute Phase Reactants in Infections: Evidence-Based Review and a Guide for Clinicians. Open Forum Infect Dis. 2015 Jul 3;2(3):ofv098. doi: 10.1093/ofid/ofv098. eCollection 2015 Sep. PMID 26258155
- [Background] Muller N, Schwarz MJ, Dehning S, Douhe A, Cerovecki A, Goldstein-Muller B, Spellmann I, Hetzel G, Maino K, Kleindienst N, Moller HJ, Arolt V, Riedel M. The cyclooxygenase-2 inhibitor celecoxib has therapeutic effects in major depression: results of a double-blind, randomized, placebo controlled, add-on pilot study to reboxetine. Mol Psychiatry. 2006 Jul;11(7):680-4. doi: 10.1038/sj.mp.4001805. Epub 2006 Feb 21. PMID 16491133
- [Background] Murray, C. J. L. et al. (1996) 'The Global burden of disease : a comprehensive assessment of mortality and disability from diseases, injuries, and risk factors in 1990 and projected to 2020 : summary / edited by Christopher J. L. Murray, Alan D. Lopez'. Geneva PP - Geneva: World Health Organization (Global burden of disease and injury series, volume 1). Available at: https://apps.who.int/iris/handle/10665/41864.
- [Background] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Background] Pizzo PA. A Prescription for Longevity in the 21st Century: Renewing Purpose, Building and Sustaining Social Engagement, and Embracing a Positive Lifestyle. JAMA. 2020 Feb 4;323(5):415-416. doi: 10.1001/jama.2019.21087. No abstract available. PMID 31917444
- [Background] Ridker PM. Clinical application of C-reactive protein for cardiovascular disease detection and prevention. Circulation. 2003 Jan 28;107(3):363-9. doi: 10.1161/01.cir.0000053730.47739.3c. No abstract available. PMID 12551853
- [Background] Tangvarasittichai S, Pongthaisong S, Tangvarasittichai O. Tumor Necrosis Factor-Alpha, Interleukin-6, C-Reactive Protein Levels and Insulin Resistance Associated with Type 2 Diabetes in Abdominal Obesity Women. Indian J Clin Biochem. 2016 Mar;31(1):68-74. doi: 10.1007/s12291-015-0514-0. Epub 2015 Jul 26. PMID 26855490
- [Background] Tipton MJ, Collier N, Massey H, Corbett J, Harper M. Cold water immersion: kill or cure? Exp Physiol. 2017 Nov 1;102(11):1335-1355. doi: 10.1113/EP086283. Epub 2017 Sep 21. PMID 28833689
- [Background] van Tulleken C, Tipton M, Massey H, Harper CM. Open water swimming as a treatment for major depressive disorder. BMJ Case Rep. 2018 Aug 21;2018:bcr2018225007. doi: 10.1136/bcr-2018-225007. PMID 30131418
- See also: The Mental Health Taskforce (2016) The Five Year Forward View For Mental Health. — https://www.england.nhs.uk/wp-content/uploads/2016/02/Mental-Health-Taskforce-FYFV-final.pdf
- See also: National Institute for Health and Care Excellence [NICE] (2018) 'Depression in adults: recognition and management [CG90]'. — https://www.nice.org.uk/guidance/cg90